CLINICAL TRIAL: NCT03989518
Title: The Link Between Mental Imagery and the Reduction of Fear in Imaginal Extinction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2019-00524
Record Dates: First submitted 2019-06-13; First posted 2019-06-18 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Healthy Subjects
Keywords: Imaginal extinction, imaginal exposure, mental imagery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simple stimuli (Experimental): Two perceptually simple stimuli are used during all experimental phases (geometrical figures).
  Interventions: Behavioral: Fear acquisition; Behavioral: Imaginal extinction; Behavioral: Reinstatement
- Complex stimuli (Experimental): Two complex stimuli are used in all experimental phases. Stimuli consist of photographs of real objects of the same size and shape as the simple stimuli, but include perceptually more complex patterns, details and colors.
  Interventions: Behavioral: Fear acquisition; Behavioral: Imaginal extinction; Behavioral: Reinstatement

INTERVENTIONS:
Behavioral: Fear acquisition — Day 1. Participants are exposed to two different visual stimuli. One of these stimuli is paired with a mild electric shock (i.e. conditioned stimuli).
Behavioral: Imaginal extinction — Day 2 (24 hours after Day 1). Participants are exposed to mental imagery of the stimuli used during fear conditioning. Imagery is prompted through different verbal instructions presented in a pseudo-randomized order. No shocks are delivered. Prior to imaginal extinction, participants receive task specific training.
Behavioral: Reinstatement — Day 3 (48 h after day1). Participants are exposed to the same stimuli used during fear conditioning (day 1) and imaginal extinction (day 2). Two unsignaled shocks are delivered at the beginning of the experiment, prior to the presentation of the first visual stimulus. No further shocks are delivered. This procedure allows the study of long term effects of imaginal extinction.

SUMMARY:
Imaginal exposure is a widely used psychological treatment technique. Imaginal extinction is an experimental analogue of imaginal exposure, that allows the study of this treatment technique under controlled circumstances (Agren, Björkstrand, & Fredrikson, 2017). During imaginal extinction, experimentally induced fear is diminished through repeated exposure to mental imagery of the feared (conditioned) stimulus. However, it is not known to what extent fear reduction depends on the mental imagery produced during this procedure. A better understanding of the mechanisms driving the effects of imaginal exposure and the factors moderating fear reduction could have significant clinical utility, by suggesting mechanistically informed ways to improve this treatment.

DETAILED DESCRIPTION:
The study takes part over three consecutive days, with fear conditioning to visual stimuli on day 1, imaginal extinction on day 2, and a fear reinstatement procedure, again to visual stimuli, on day 3. Skin conductance is used to measure fear responses.

Participants' are randomized to receive conditioning, extinction and reinstatement with either complex or simple stimuli. During imaginal extinction, imagery of each experimental stimulus is prompted through different verbal instructions.

ELIGIBILITY:
Inclusion Criteria:

Age 18 or over

Fluent in Swedish

Willing and able to provide informed consent and complete study procedures

Exclusion Criteria:

Current psychiatric disorder

Use of psychotropic medication within 6 months prior to study start

Receiving psychological treatment within 6 months prior to study start

Current neurological condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Skin conductance response (SCR) | Day 1
  SCR is used as a measure of physiological fear responses. Differences in fear responses are used to assess fear learning during fear acquisition and to explore main effects and interactions between fear learning, stimulus complexity and capacity for mental imagery.
Skin conductance response (SCR) | Day 2 (24 h after day1)
  SCR is used as a measure of physiological fear responses.Differences in fear responses are used to assess fear reduction during imaginal extinction, and to explore main effects and interactions between fear reduction, stimulus complexity and capacity for mental imagery.
Skin conductance response (SCR) | Day 3 (48 h after day 1)
  SCR is used as a measure of physiological fear responses.Differences in fear response are used to assess return of fear during reinstatement, and to explore main effects and interactions between return of fear, stimulus complexity and capacity for mental imagery.

SECONDARY OUTCOMES:
Fear ratings | Day 1
  Ratings of subjective fear during the experimental procedure. Scale: 0 -100 (no fear at all - extreme fear)
State-Trait Anxiety Inventory | Day 1
  This is a self-rated questionnaire measuring trait anxiety. Higher scores indicate higher level of trait-anxiety (range 20-80)
Difficulties in emotion regulation scale | Day 1
  This is a self-rated questionnaire measuring difficulties in emotion regulation. Higher scores indicate higher level of difficulties in emotion regulation (range 36-180)
Fear ratings | Day 2 (24 h after day 1)
  Ratings of subjective fear during the experimental procedure. Scale: 0 -100 (no fear at all - extreme fear)
Vividness of mental imagery during imaginal extinction | Day 2 (24 h after day 1)
  Scale: 1-5; no image at all - image as clear and vivid as real life
The Plymouth Sensory Imagery Questionnaire | Day 2 (24 h after day 1)
  This is a self-rated questionnaire measuring vividness of mental imagery across different sensory modalities. Higher scores indicate higher level of vividness. (range 0-70)
The Vividness of Visual Imagery Questionnaire | Day 2 (24 h after day 1)
  This is a self-rated questionnaire measuring vividness of visual mental imagery. Only eyes open section is administered. Higher scores indicate higher level of vividness (range 0-80)
Spontaneous use of imagery scale | Day 2 (24 h after day 1)
  This is a self-rated questionnaire measuring spontaneous use of imagery. Higher scores higher levels use of spontaneous use of imagery (range 12- 60)
Expectancy ratings | Day 2 (24 h after day 1)
  After the imaginal extinction procedure, participants are asked to rate to what extent they believed that electric shocks would be delivered during the procedure on a scale ranging from 0 - 100 %
Fear ratings | Day 3 (48 h after day 1)
  Ratings of subjective fear during the experimental procedure. Scale: 0 -100 (no fear at all - extreme fear)
Expectancy ratings | Day 3 (48 h after day 1)
  After the reinstatement procedure, participants are asked to rate to what extent they believed that electric shocks would be delivered during the procedure on a scale ranging from 0 - 100 %

OTHER OUTCOMES:
Task compliance | Day 1
  Questions asking participants to rate to what extent they followed the instructions during the experimental procedure on a scale ranging from 0 - 100 %.
Task compliance | Day 2 (24 h after day 1)
  Questions asking participants to rate to what extent they followed the instructions during the experimental procedure on a scale ranging from 0 - 100 %.
Task compliance | Day 3 (48 h after day 1)
  Questions asking participants to rate to what extent they followed the instructions during the experimental procedure on a scale ranging from 0 - 100 %.

CONTACTS AND LOCATIONS:
Locations (1):
- Uppsala University, Departement of Psychology, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available upon publication.

REFERENCES:
- [Background] Agren T, Bjorkstrand J, Fredrikson M. Disruption of human fear reconsolidation using imaginal and in vivo extinction. Behav Brain Res. 2017 Feb 15;319:9-15. doi: 10.1016/j.bbr.2016.11.014. Epub 2016 Nov 10. PMID 27840245